CLINICAL TRIAL: NCT01963988
Title: Pilot Study for Comparison of the Efficacy Between Transurethral Coagulation and Transurethral Resection of Ulcer in Bladder Pain Syndrome Patients
Brief Title: Comparison of the Efficacy Between Transurethral Coagulation and Transurethral Resection of Ulcer in Bladder Pain Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor,MD,PhD, Samsung Medical Center
Other Study IDs: 2013-05-127; ksleedr (Registry Identifier: LKS)
Record Dates: First submitted 2013-07-15; First posted 2013-10-17 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Bladder Pain Syndrome
Keywords: Bladder Pain Syndrome; Transurethral Resection of Ulcer; Transurethral Coagulation of Ulcer
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transurethral Coagulation (TUC): This cohort patients will be managed with Transurethral Coagulation (TUC) of IC ulcer lesion
  Interventions: Procedure: Transurethral Coagulation (TUC)
- Transurethral Resection(TUR): This cohort patients will be managed with transurethral resection(TUR) of IC ulcer lesion
  Interventions: Procedure: Transurethral Resection(TUR)

INTERVENTIONS:
Procedure: Transurethral Coagulation (TUC)
  Groups: Transurethral Coagulation (TUC)
Procedure: Transurethral Resection(TUR)
  Groups: Transurethral Resection(TUR)

SUMMARY:
On the EAU (European Association of Urology) guidelines, the ulcer type bladder pain syndrome (BPS) should be treated with transurethral resection (TUR) or coagulation (TUC) of ulcer.

But, Up to date, there was no study to compare the therapeutic efficacy of TUR with TUC in ulcer type BPS patients.

We assume TUR have a more therapeutic effect than TUC.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 yrs or greater
2. Patients diagnosed with BPS(Bladder Pain Syndrome)
3. Symptom persisted more than 6 months
4. Pain VAS ≥4
5. O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) scores 12 or greater with pain and nocturia domain scores > 2.
6. Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF) >13
7. No history of cystoscopy within 2yrs.

Exclusion Criteria:

1. History of augmentation cystoplasty or previous transurethral coagulation/resection due to BPS
2. Child-bearing potential, pregnant or nursing women.
3. Mean voided volume lesser than 40ml or over than 400ml.
4. Hematuria exceeds 1+ in the urinary dipstick (dipstick) examination.
5. Urinary tract infection during run-in periods.
6. Genitourinary tuberculosis or bladder,urethral and prostate cancer
7. Recurrent urinary tract infection
8. History of hysterectomy,mid-urethral sling,pelvic organ prolapse repair,vaginal delivery or Cesarean section,prostate operation or treatment etc within 6months.
9. Neurologic disease history of cerebral infarction,multiple sclerosis or parkinsonism etc.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled diagnosed with bladder pain syndrome by ESSIC proposal.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival between TUC and TUR | Until 12 months after the last subject be enrolled

SECONDARY OUTCOMES:
The change of voiding dairy parameters(mean number of micturition,Urgency etc) after each treatment | 1,3,6,9 and 12 months
The change of Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF) | 1,3,6,9 and 12months.
The change of Global Response Assessment(GRA) score | 1,3,6,9 and 12 months
The change of EQ-5D (EuroQOL five dimensions) Health Questionnaire score | 1,3,6,9 and 12months
The change of Patient Global Assessment(PGA) | 12months
The change of Brief Pain Inventory-short form(BPI-sf) score | 9 and 12months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea